CLINICAL TRIAL: NCT02850172
Title: Effects of a "Walk, Eat, & Breathe" Nursing Intervention For Patients With Esophageal Cancer: A Randomized Controlled Trial
Brief Title: Effects of a "Walk, Eat, & Breathe" Nursing Intervention For Patients With Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201602045RINC
Record Dates: First submitted 2016-05-11; First posted 2016-07-29 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Esophageal Cancer
Keywords: nutrition; exercise; inspiratory muscle training
MeSH Terms: conditions — Esophageal Neoplasms; Motor Activity | interventions — Walking; Eating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walk, eat, & breathe group (Experimental): Participants in the experimental group will receive "Walk, Eat, & Breathe" at initiation of CCRT and ends before curative surgery.
  Interventions: Behavioral: Walk, Eat, & Breathe
- Control group (No Intervention): Participants in the control group received usual care.

INTERVENTIONS:
Behavioral: Walk, Eat, & Breathe — 1. Walking exercise: 3 times per week, 20~30 mins per section
  2. Eat: nutritional assessment and advice weekly
  3. Inspiratory muscle training: twice every day, 7 days a week, 6~8 weeks before surgery
  Arms: Walk, eat, & breathe group

SUMMARY:
The purpose of this stratified randomized controlled trial (RCT) is to test the effects of Walk, Eat, & Breathe on preserving patients' nutritional status, functional walking capacity, pulmonary function, and emotional well-being during the CCRT and surgery course.Additionally, effects to reduce treatment-related complications and length of hospital stay for esophagectomy will be evaluated between experimental and control groups.

DETAILED DESCRIPTION:
Esophageal cancer is a devastating disease with poor prognosis. This is largely due to its rather insidious progression, so most patients were diagnosed with advanced cancer stage. Patients with advanced stage therefore have to be treated with neoadjuvant chemoradiotherapy (CCRT) to shrink the tumor and followed by a curative surgery (i.e., esophagectomy). Patients' nutritional status, functional walking capacity, and emotional well-being are substantially deteriorated, which often increase the incidence of postoperative pulmonary complications, thus the risk of surgical death is greatly increased. To better support patients with esophageal cancer, during this critical treatment course (approximate 4 months in length), we develop a "Walk, Eat, & Breathe" nursing intervention consisting of nutritional advice, walking exercise, and inspiratory muscle training. The purpose of this stratified randomized controlled trial (RCT) is to test the effects of Walk, Eat, & Breathe on preserving patients' nutritional status, functional walking capacity, pulmonary function, and emotional well-being during the CCRT and surgery course. Additionally, effects to reduce treatment-related complications and length of hospital stay for esophagectomy will be evaluated between experimental and control groups.

For this three-year stratified RCT, a total of 144 consecutive patients will be enrolled to ensure the power of study. Patients will be eligible for the study if they had histologically documented, locally advanced tumors of the esophagus, defined as American Joint Committee on Cancer (AJCC) stage IIB or higher, were scheduled for neoadjuvant chemoradiotherapy and subsequent curative surgery, and had no contraindication precluding walking. After obtaining the consent, participants will be first stratified by two important covariates [intake status (oral intake or tube feeding) and tumor location (upper third or middle & lower third of esophagus)] and then randomized separately into the experimental or control group, according to computer-generated randomization tables.

Participants in the experimental group will receive "Walk, Eat, & Breathe" at initiation of CCRT and ends before curative surgery. Participants in the control group received usual care. Participants will undergo measurements at four points in time: before CCRT, after CCRT, before surgery, and 1-month after surgery. Primary endpoints include nutritional status (body weight, lean muscle mass), functional walking capacity (hand-grip strength, 6-min walking distance), pulmonary function (forced vital capacity, forced expiratory volume in 1 second, maximal inspiratory pressure), and emotional well-being (anxiety/depression, quality of life). Secondary endpoints include treatment-related complications and length of hospital stay for esophagectomy. The treatment-related complications will include chemoradiotherapy-related toxicity (i.e., neutropenia, esophagitis), rates of interruptions (i.e., discontinuation, reduction) in chemotherapy or radiotherapy, unplanned hospital admission, incidence of postoperative pulmonary complications, and length of mechanical ventilation for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. the patient is cognitively capable to understand the trial;
2. locally advanced tumors of the esophagus, defined as American Joint Committee on Cancer (AJCC) stage IIB or higher, were scheduled for neoadjuvant chemoradiotherapy and subsequent curative surgery;
3. the patient is willing to sign the informed consent form.

Exclusion Criteria:

1. age <20 years;
2. the patient is unable to communicate in the Chinese language; and
3. the patient has contraindications that limit physical activity such as severe cardiac disease, recent myocardial infarction or uncontrolled hypertension.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Body weight | 5 months
  Record the trajectory of body weight during cancer treatment
Lean muscle mass | 5 months
  Record the trajectory of lean muscle mass during cancer treatment using bioelectrical impedance analysis
functional walking capacity | 5 months
  Record the trajectory of walking capacity during cancer treatment using 6-min walk test
hand-grip strength | 5 months
  Record the trajectory of hand-grip strength during cancer treatment using Hand-held dynamometer
pulmonary function | 5 months
  Record the trajectory of pulmonary function(FVC, FEV1) during cancer treatment using spirometry. The parameters are recorded with the prediction values of FVC% and FEV1%.
maximal inspiratory pressure | 5 months
  Record the trajectory of maximal inspiratory pressure during cancer treatment using inspiratory training device: POWERbreathe KH1
anxiety and depression (HADS questionnaire) | 5 months
  Record the trajectory of anxiety and depression during cancer treatment
quality of life (EORTC-QLQ-C30 questionnaire) | 5 months
  Record the trajectory of quality of life during cancer treatment
severity of symptom (QLQ-OES18 questionnaire) | 5 months
  Record the trajectory of severity of symptom during cancer treatment

SECONDARY OUTCOMES:
chemoradiotherapy-related toxicity (CTCAE grading system) | 5 months
  Record the severity of chemoradiotherapy-related toxicity during cancer treatment
length of hospital stay | 5 months
  Record the length of hospital stay for esophagectomy
treatment interruptions | 5 months
  Record the "event" of treatment discontinuation or reduction on chemotherapy or radiotherapy. The result was coded as "yes" or "no". The variable are depicted in term of frequency and percentage of participants with treatment interruptions during cancer treatment
unplanned hospital admission | 5 months
  Record the "event" of unplanned hospital admission. The result was coded as "yes" or "no". The variable are depicted in term of frequency and percentage of participants with unplanned hospital admission during cancer treatment
postoperative pulmonary complications | 30 days
  Record the incidence of postoperative pulmonary complications included pneumonia, acute respiratory distress syndrome (ARDS) and respiratory insufficiency developing within 30 days after surgery
length of mechanical ventilation | 30 days
  Record the length of mechanical ventilation after esophagectomy (coded as hours)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Chia-Hui Chen, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided